CLINICAL TRIAL: NCT02929316
Title: Vedolizumab Induction May Prevent Celiac Enteritis After Gluten Challenge in Established Celiac Patients in Histological Remission
Brief Title: Vedolizumab Induction May Prevent Celiac Enteritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: AGA Clinical Research Associates, LLC (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Barry Kaufman, MD, Director of Clinical Research, AGA Clinical Research Associates, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IISR-2016-101481
Record Dates: First submitted 2016-10-05; First posted 2016-10-11 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vedolizumab (Experimental): Vedolizumab (Entyvio) 300mg IV at week 0, 2 and 6
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — IV infusion week 0, 2 and 6
  Other Names: Entyvio

SUMMARY:
Celiac disease (CD) is characterized as an autoimmune disorder whereby gluten (a protein found in wheat, barley, rye, malt) induces an immunological response in genetically susceptible individuals. The prevalence of CD has been estimated to affect 0.5-1% of the population worldwide. Long term sequelae are numerous and include risk of lymphoma, malabsorption leading to weight loss, anemia, multiple vitamin deficiencies, osteoporosis/osteopenia, secondary autoimmunity, etc. (1)

DETAILED DESCRIPTION:
Adult subjects with CD will be recruited through our clinic. All patients enrolled will have established CD diagnosed > 6 months. All patients will have history of abnormal MARSH score on initial duodenal biopsy at diagnosis and MARSH 0 on repeat biopsy following a gluten free diet (GFD). All patients will also have positive celiac serologies (anti-TTG, anti-gliadin, etc.) at diagnosis, as well as, positive HLA DQ2/DQ8 genetic profile. At enrollment, all patients will have negative celiac serologies, indicative of serologic remission on a gluten free diet. Female subjects of childbearing potential (does not include those with history of tubal ligation/surgical sterilization, hysterectomy and/or oophorectomy) who are sexually active with a non-sterilized male partners agree to routinely use adequate contraception from signing informed consent, during study process and for an additional 18 weeks after the last dose of vedolizumab. A male subject who is non-sterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing informed consent throughout the duration of the study and for 18 weeks after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following criteria for study entry:
* Adult patients with Celiac Disease (CD)
* Without any additional co-morbidities
* Normal renal and hepatic function
* Diagnosis of CD established at least 6 months prior to trial with diagnostic serology, genetic profile, endoscopic appearance and histopathology report In histologic and serologic remission (defined as MARSH 0 and negative anti-tissue transglutaminase, etc.) following a gluten free diet
* Naïve to treatment with vedolizumab
* Able and willing to provide written informed consent
* Eligibility criteria for laboratory profiles - healthy patient normal laboratory reference values

  * WBC 4.5-12.0 k/UL
  * Platelet count- 140-415 k/UL
  * Hemoglobin- 11.0-17.4 %g/dL
  * Renal Function-
  * Creatinine- 0.5-1.3 mg/dL
  * BUN- 5-20 mg/dL
  * Hepatic Function
  * Albumin - 3.3-5.0 g/dL
  * INR- 0.9-1.1
  * AST- 0-37 U/L
  * ALT- 0-40 U/L
  * Total Bilirubin- 0.1-1.3 mg/dL
  * Alk Phos- 35-150 U/L

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from study entry:
* Abnormal MARSH score on enrollment histopathology
* Elevated celiac serologies (anti-tissue transglutaminase, etc.)
* Current use of biologics or immunomodulators Adalimumab, infliximab, Ustekinumab, Golimumab, Tocilizumab, Certolizumab, Etanercept, Rituximab, Anakinra, Abatacept, Tofacitinib, Methotrexate, Azathioprine, 6-MP.
* Current use of immunosuppressive therapy including intermittent systemic corticosteroids within two months of vedolizumab induction
* History of intestinal lymphoma (MALToma, etc.)
* History of cancer including hematologic malignancy, solid tumors, carcinoma in situ, etc.
* Pregnant or lactating
* Fertile females will require at least one form of birth control
* Lack of peripheral venous access
* Inability to comply with study protocol, in the opinion of the investigator
* Neurological conditions which may interfere with monitoring for PML
* History of demyelinating disease or history of major neurological disease
* History of alcohol, drug or chemical abuse < 6 months prior to screening
* History of active tuberculosis (TB) or a positive screening test for latent mycobacterium tuberculosis infection
* Positive PPD= > 10 mm or > 5mm in patients on 15 mg or more of prednisone
* History of BCG vaccination should be screened using Quantiferon TB Gold test
* An Indeterminate Quantiferon test will require a chest X-ray to rule out active TB and consultation with an infectious disease specialist to confirm the risk of latent
* TB is low and that patients can be safely enrolled in the trial
* History of recurrent opportunistic infections and/or of severe or disseminated viral infections
* Active autoimmune disease
* Active inflammatory bowel disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Normal histopathology following induction dosing with vedolizumab | 12 weeks
  Remission is defined in this study of negative celiac antibodies and normal duodenal biopsies
Normal histopathology following induction dosing with vedolizumab after 2 week gluten challange | 12 weeks
  Remission is defined in this study as negative celiac antibodies and normal duodenal biopsies

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - Theresa Stevens, Egg Harbor, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Green PH, Cellier C. Celiac disease. N Engl J Med. 2007 Oct 25;357(17):1731-43. doi: 10.1056/NEJMra071600. No abstract available. PMID 17960014
- [Result] Lionetti E, Castellaneta S, Francavilla R, Pulvirenti A, Tonutti E, Amarri S, Barbato M, Barbera C, Barera G, Bellantoni A, Castellano E, Guariso G, Limongelli MG, Pellegrino S, Polloni C, Ughi C, Zuin G, Fasano A, Catassi C; SIGENP (Italian Society of Pediatric Gastroenterology, Hepatology, and Nutrition) Working Group on Weaning and CD Risk. Introduction of gluten, HLA status, and the risk of celiac disease in children. N Engl J Med. 2014 Oct 2;371(14):1295-303. doi: 10.1056/NEJMoa1400697. PMID 25271602
- [Result] Lee SK, Lo W, Memeo L, Rotterdam H, Green PH. Duodenal histology in patients with celiac disease after treatment with a gluten-free diet. Gastrointest Endosc. 2003 Feb;57(2):187-91. doi: 10.1067/mge.2003.54. PMID 12556782
- [Result] Leffler DA, Schuppan D. Update on serologic testing in celiac disease. Am J Gastroenterol. 2010 Dec;105(12):2520-4. doi: 10.1038/ajg.2010.276. PMID 21131921
- [Result] Wahab PJ, Meijer JW, Mulder CJ. Histologic follow-up of people with celiac disease on a gluten-free diet: slow and incomplete recovery. Am J Clin Pathol. 2002 Sep;118(3):459-63. doi: 10.1309/EVXT-851X-WHLC-RLX9. PMID 12219789
- [Result] Vahedi K, Mascart F, Mary JY, Laberenne JE, Bouhnik Y, Morin MC, Ocmant A, Velly C, Colombel JF, Matuchansky C. Reliability of antitransglutaminase antibodies as predictors of gluten-free diet compliance in adult celiac disease. Am J Gastroenterol. 2003 May;98(5):1079-87. doi: 10.1111/j.1572-0241.2003.07284.x. PMID 12809831
- [Result] Kelly CP, Green PH, Murray JA, Dimarino A, Colatrella A, Leffler DA, Alexander T, Arsenescu R, Leon F, Jiang JG, Arterburn LA, Paterson BM, Fedorak RN; Larazotide Acetate Celiac Disease Study Group. Larazotide acetate in patients with coeliac disease undergoing a gluten challenge: a randomised placebo-controlled study. Aliment Pharmacol Ther. 2013 Jan;37(2):252-62. doi: 10.1111/apt.12147. Epub 2012 Nov 19. PMID 23163616
- [Result] Leffler DA, Kelly CP, Abdallah HZ, Colatrella AM, Harris LA, Leon F, Arterburn LA, Paterson BM, Lan ZH, Murray JA. A randomized, double-blind study of larazotide acetate to prevent the activation of celiac disease during gluten challenge. Am J Gastroenterol. 2012 Oct;107(10):1554-62. doi: 10.1038/ajg.2012.211. Epub 2012 Jul 24. PMID 22825365
- [Result] Leffler D, Schuppan D, Pallav K, Najarian R, Goldsmith JD, Hansen J, Kabbani T, Dennis M, Kelly CP. Kinetics of the histological, serological and symptomatic responses to gluten challenge in adults with coeliac disease. Gut. 2013 Jul;62(7):996-1004. doi: 10.1136/gutjnl-2012-302196. Epub 2012 May 22. PMID 22619366